CLINICAL TRIAL: NCT01993823
Title: A Phase III, Multicenter, Randomized, Double-blind, Parallel Group, Active Treatment-controlled Study Assessing the Safety and Efficacy of G238 Compared to Clotrimazole 1% Otic Solution in Patients With Otomycosis
Brief Title: Clinical Study to Assess the Efficacy and Safety of G238 Compared to Clotrimazole Otic Solution in the Treatment of Otomycosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Salvat (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G238OTIII/11IA01
Record Dates: First submitted 2013-10-09; First posted 2013-11-25 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Otomycosis
MeSH Terms: conditions — Otomycosis | interventions — Clotrimazole

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- G238 (Experimental): Five drops into the ear canal twice daily for 14 days
  Interventions: Drug: G238
- Clotrimazole (Active Comparator): Five drops into the ear canal twice daily for 14 days
  Interventions: Drug: Clotrimazole

INTERVENTIONS:
Drug: G238 — Five drops into the ear canal twice daily for 14 days
  Arms: G238
Drug: Clotrimazole — Five drops into the ear canal twice daily for 14 days
  Arms: Clotrimazole

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of G238 for the treatment of otomycosis

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Clinical diagnosis of otomycosis where topical treatment is indicated.

Exclusion Criteria:

* Other ear diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratorios SALVAT, S.A., Esplugues de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Lee A, Tysome JR, Saeed SR. Topical azole treatments for otomycosis. Cochrane Database Syst Rev. 2021 May 25;5(5):CD009289. doi: 10.1002/14651858.CD009289.pub2. PMID 34033120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: ENT Mexican sites
Period: Overall Study
Arm/Group | G238 | Clotrimazole
Started | 95 | 95
Completed | 88 | 79
Not Completed | 7 | 16
Not completed — Requested by the patient | 6 | 11
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Population: ITT population: Randomized patients who had at least one efficacy evaluation after starting treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | G238 | Clotrimazole | Total
Number analyzed (Participants) | 89 | 85 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (15.8) | 39.8 (13.0) | 40.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 46 | 90
  Male | 45 | 39 | 84

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With a Complete Response to Treatment
Description: Efficacy will be assessed primarily by evaluation of the fungal culture, and the sum of signs and symptom scores (pruritus, otalgia, otorrhea and aural fullness obstruction to be scored as 0=absent; 1= mild; 2=moderate; 3=severe). The primary efficacy variable is the proportion of subjects with a negative culture for fungus, AND a signs and symptom score of 0 on Day 24.
  Response to the study treatment was classed according to the following definitions:
  * Complete response: Negative fungal culture or presumed eradication on day 24, and sum score for signs and symptoms = 0 on day 24.
  * Partial response: Negative culture or presumed eradication on day 24, and sum score for signs and symptoms = 1 or 2 on day 24.
  * No response: Positive culture on day 24 or negative culture or presumed eradication and sum score for signs and symptoms > 2 on day 24.
Time Frame: Day 24
Population: ITT
Measure: Number; unit: participants
Arm/Group | G238 | Clotrimazole
Number analyzed (Participants) | 89 | 85
participants
  Complete Response | 72 | 66
  Partial Response | 11 | 11
  No-response | 5 | 2
  Missing data | 1 | 6

2. Secondary Outcome: Changes in Signs/ Symptoms
Description: The secondary efficacy variables include:
  * Proportion of subjects with signs and symptoms score of "0" at Day 15
  * Proportion of subjects with signs and symptoms score of "0" at Day 24
  * Proportion of subjects with a negative culture for fungus or presumed eradication (mycological cure) on Day 24.
Time Frame: 2 weeks and 4 weeks
Population: ITT
Measure: Number; unit: percentage of patient
Arm/Group | G238 | Clotrimazole
Number analyzed (Participants) | 89 | 85
percentage of patient
  Signs and symptoms score 0 at Day 15 | 59.55 | 77.65
  Signs and symptoms score 0 at Day 24 | 85.83 | 86.08
  Mycological cure at Day 24 | 96.63 | 97.65

3. Other Pre Specified Outcome: Mycological Study
Time Frame: Day 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The safety analysis was conducted on the safety population (SAF), i.e. the population that includes all the randomised subjects who took at least one dose of the trial drug and had a safety evaluation.
Arm/Group | G238 | Clotrimazole
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/85
Other Adverse Events (participants affected / at risk) | 0/89 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor does not object to publication by Institution of the results of the Trial based on information collected or generated by Institution, whether or not the results are favorable to the Sponsor Drug. However, to ensure against inadvertent disclosure of Confidential Information or unprotected Inventions, Institution will provide Sponsor an opportunity to review any proposed publication or other type of disclosure before it is submitted or otherwise disclosed.